CLINICAL TRIAL: NCT03193853
Title: Phase II Clinical Trial of Treatment With TAK-228 and TAK-117 to Inhibit Homologous Recombination (HR) Followed by Cisplatin and Nab Paclitaxel in Patients With Chemotherapy-pretreated Metastatic Triple Negative Breast Cancer
Brief Title: TAK-228 and TAK-117 Followed by Cisplatin and Nab Paclitaxel for Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joyce O'Shaughnessy (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Joyce O'Shaughnessy, Medical Oncologist/Medical Director, Baylor Research Institute
Organization: Baylor Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017- 113; Baylor 017-113 (Other: Baylor Scott & White Research Institute)
Record Dates: First submitted 2017-06-09; First posted 2017-06-21 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sapanisertib; serabelisib; Cisplatin; Taxes

STUDY DESIGN:
Intervention Model Description: Patients with metastatic TNBC who meet the enrollment criteria will receive TAK-228 and TAK-117 until disease progression followed by nab paclitaxel plus cisplatin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tak + cisplatin and nab paclitaxel (Experimental): Patients with metastatic TNBC who meet the enrollment criteria will receive TAK-228 and TAK-117 until disease progression followed by nab paclitaxel plus cisplatin for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion.
  Interventions: Drug: Tak-228 & Tak-117; Drug: Cisplatin & Nab Paclitaxel

INTERVENTIONS:
Drug: Tak-228 & Tak-117 — Patients will receive 4mg oral TAK-228 and 200mg TAK-117 tablets until disease progression.
Drug: Cisplatin & Nab Paclitaxel — following Tak-228 & Tak-117 standard nab paclitaxel 175-220 mg/m2 plus cisplatin 60-75 mg/m2 infusion for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion

SUMMARY:
This study evaluates efficacy of TAK- 228 and TAK- 117 followed by cisplatin and nab paclitaxel in patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
Seventy to eighty percent of breast cancers have a gene expression profile which is characterized by homologous recombination deficiency (HRD) and high proliferation. HRD leads to errors in DNA pathway [non -homologous end joining (NHEJ)] that repair DNA-breaks, a process required for metastatic triple negative breast cancer (TNBC) survival. The hypothesis of this pilot trial is that administration of the oral combination of TAK-228 and TAK-117 (PIKTOR) will inhibit NHEJ in metastatic TNBC, leading at the time of disease progression to metastases that are HR-deficient and sensitive to cisplatin plus nab paclitaxel therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years or older.
2. Have a diagnosis of metastatic TNBC previously treated with standard anthracycline, cyclophosphamide, and taxane chemotherapy, unless there was a contraindication to doxorubicin, in which case prior treatment with this agent is not required.
3. Have not received more than 3 prior chemotherapy regimens for metastatic disease. Prior platinum and/or taxane therapy in the adjuvant or metastatic setting is permitted.
4. Androgen receptor-negative (less than 10% positive nuclei) on standard IHC performed at the local pathology laboratory.
5. Have locoregional (eg, breast, chest wall, regional lymphatic) or pulmonary or hepatic metastatic disease that is amenable to core needle biopsy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (See Appendix I)
7. Female patients who:

   1. Are postmenopausal for at least 1 year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential, agree to practice 1 effective methods of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer as mandated by local labeling [eg, USPI, SmPC, etc,]) after the last dose of study drug, OR
   4. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
8. Screening clinical laboratory values as specified below:

   1. Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥ 1.5 x 10^9; platelet count ≥ 100 x 10^9; hemoglobin ≥ 9 g/dL without transfusion within 1 week preceding study drug administration
   2. Hepatic: total bilirubin ≤ 1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase-AST/SGOT and alanine aminotransferase/serum glutamic pyruvic transaminase-ALT/SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present);
   3. Renal: creatinine clearance ≥60 mL/min based either on cockroft-Gault estimate or based on urine collection (12 or 24 hour);
   4. Metabolic: Glycosylated hemoglobin (HbA1c)<7.0%, fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL
9. Ability to swallow oral medications.
10. Must be able to fast for glucose monitoring throughout PIKTOR treatment.
11. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

    1. Brain metastases which have been treated
    2. No evidence of disease progression for ≥2 months before the first dose of study drug.
    3. No hemorrhage after treatment
    4. Off-treatment with dexamethasone for 3 weeks before administration of the first dose of PIKTOR
    5. No ongoing requirement for dexamethasone or anti-epileptic drugs
12. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Leptomeningeal disease that is symptomatic or cytology-proven.
2. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study.
3. Known human immunodeficiency virus infection.
4. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
6. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
7. Breast feeding or pregnant.
8. Treatment with any investigational products within 30 days before the first dose of study drug
9. Previous treatment with PI3K, AKT, dual PI3K/mTOR inhibitors, TORC1/2 inhibitors or TORC1 inhibitors.
10. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of PIKTOR. In addition, patients with enteric stomata are also excluded.
11. History of any of the following within the last 6 months before administration of the first dose of the drug:

    1. Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
    2. Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
    3. Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
    4. Placement of a pacemaker for control of rhythm
    5. New York Heart Association (NYHA) Class III or IV heart failure f. Pulmonary embolism
12. Significant active cardiovascular or pulmonary disease including:

    1. Uncontrolled hypertension (ie, systolic blood pressure >180 mm Hg, diastolic blood pressure > 100 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle1 Day 1 is allowed.
    2. Pulmonary hypertension
    3. Need for supplemental oxygen
    4. Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
    5. Medically significant (symptomatic) bradycardia
    6. History of arrhythmia requiring an implantable cardiac defibrillator
    7. Baseline prolongation of the rate-corrected QT interval (QTc) (eg, repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes)
13. Poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) > 7%; patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met.
14. Treatment with strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4, CYP2C19 or CYP2C19 within 1 week preceding the first dose of study drug (See Appendix IV).
15. Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy) within 1 week before administration of the first dose of study drug.
16. Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Patients
Enrollment: 12 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — Baylor Scott & White Research Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Investigators will share de-identified data with Takeda for information/publication purposes

REFERENCES:
- [Derived] Lang JD, Nguyen TVV, Levin MK, Blas PE, Williams HL, Rodriguez ESR, Briones N, Mueller C, Selleck W, Moore S, Zismann VL, Hendricks WPD, Espina V, O'Shaughnessy J. Pilot clinical trial and phenotypic analysis in chemotherapy-pretreated, metastatic triple-negative breast cancer patients treated with oral TAK-228 and TAK-117 (PIKTOR) to increase DNA damage repair deficiency followed by cisplatin and nab paclitaxel. Biomark Res. 2023 Jul 25;11(1):73. doi: 10.1186/s40364-023-00511-7. PMID 37491309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients are not included in the results as they screen failed before begin assigned to a study group.
Groups:
- Tak + Cisplatin and Nab Paclitaxel: Patients with metastatic TNBC who meet the enrollment criteria will receive TAK-228 and TAK-117 until disease progression followed by nab paclitaxel plus cisplatin for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion.
  Tak-228 & Tak-117: Patients will receive 4mg oral TAK-228 and 200mg oral TAK-117 tablets until disease progression.
  Cisplatin & Nab Paclitaxel: following Tak-228 & Tak-117 standard 175-220 mg/m2 nab paclitaxel plus 60-75 mg/m2 cisplatin infusion for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion
Period: Overall Study
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Started | 10
Completed | 4
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Groups:
- Tak + Cisplatin and Nab Paclitaxel: Patients with metastatic TNBC who meet the enrollment criteria will receive TAK-228 and TAK-117 until disease progression followed by nab paclitaxel plus cisplatin for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion.
  Tak-228 & Tak-117: Patients will receive oral TAK-228 and TAK-117 tablets until disease progression.
  Cisplatin & Nab Paclitaxel: following Tak-228 & Tak-117 standard nab paclitaxel plus cisplatin infusion for six cycles. Patients who did not progress may continue nab paclitaxel under treating physicians discretion
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 52 [41 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Objective Response Rate)
Description: To assess the objective response rate associated with sequential treatment of the oral combination TAK 228 and 117 followed by nab-paclitaxel plus cisplatin in metastatic TNBC. Objective response is measured as prolonged clinical benefit; clinical benefit is defined as progression free survival on study therapy for at least 6 months.
Time Frame: Through study completion, up to 2 years 8 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Number analyzed (Participants) | 10
Participants | 1

2. Secondary Outcome: Efficacy (Duration of Response)
Description: To assess duration of response associated with sequential treatment of the oral combination Tak 228 and 117 followed by nab-paclitaxel plus cisplatin. Duration of response is measured as prolonged clinical benefit; clinical benefit is defines as progression free survival on study therapy for at least 6 months.
Time Frame: Through study completion, up to 2 years 8 months
Measure: Number; unit: weeks
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Number analyzed (Participants) | 1
weeks | 28

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0".
Description: To assess safety associated with sequential treatment of the oral combination Tak 228 and 117 followed by nab-paclitaxel plus cisplatin
Time Frame: For up to 30 days following last dose, approximately 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: Number of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: To assess safety associated with sequential treatment of the oral combination TAK 228 and TAK 117 followed by nab-paclitaxel plus cisplatin per CTCAE v4.0 criteria.
Time Frame: For up to 30 days following last dose, approximately 7 months
Measure: Number; unit: adverse events
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
Number analyzed (Participants) | 10
adverse events | 64

ADVERSE EVENTS:
Time Frame: For up to 30 days following last dose, approximately 7 months
Description: All AEs are recorded for up to 30 days following the last dose of study treatment, approximately 7 months
Arm/Group | Tak + Cisplatin and Nab Paclitaxel
All-Cause Mortality (participants affected / at risk) | 6/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tak + Cisplatin and Nab Paclitaxel (N=10)
Renal Injury (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transient ischemic attack (Vascular disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tak + Cisplatin and Nab Paclitaxel (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Axilla Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bacterial Vaginosis (Infections and infestations) | 1 (1)
Blurred Vision (General disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cervicalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Decreased Appetite (General disorders) | 1 (1)
Dehydration (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dizziness (General disorders) | 3 (3)
Dry Throat (General disorders) | 1 (1)
Dysgeusia (General disorders) | 2 (2)
Dysphagia (General disorders) | 1 (1)
Dysphonia (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Earache (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 4 (5)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hoarseness (General disorders) | 2 (2)
Hot Flashes (General disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 3 (3)
Hyperopia (General disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Ictericia (Hepatobiliary disorders) | 1 (1)
Increased Forgetfulness (General disorders) | 1 (1)
Insomnia (General disorders) | 3 (3)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 3 (3)
Lethargy (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (10)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2)
Neuropathy in Lower Extremities (Nervous system disorders) | 5 (5)
Neuropathy in Upper Extremities (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Scalp Tenderness (Skin and subcutaneous tissue disorders) | 1 (1)
Shin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore Throat (Infections and infestations) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Strep Throat (Infections and infestations) | 2 (2)
Thrombus (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Transaminitis (Hepatobiliary disorders) | 2 (2)
Tremors (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3)
Viral Gastroenteritis (Infections and infestations) | 1 (1)
Vision Changes (Eye disorders) | 1 (1)
Vitamin D Deficiency (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03193853/Prot_SAP_000.pdf